CLINICAL TRIAL: NCT03855488
Title: Imagery Enhanced Cognitive Bias Modification for Chronic Worry
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: No in-person testing is permitted at Ryerson University due to COVID-19.
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Ministry of Research, Innovation and Science, Ontario (Other)
Responsible Party: Principal Investigator, Bailee Malivoire, PhD Student, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 2018-394
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Excessive Worry
Keywords: Worry; Anxiety; Imagery; Cognitive bias modification
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Baseline (pre-intervention) outcome measures will be completed at the first visit to our lab at Ryerson University. Participants will then be randomly assigned to one of the following conditions: (1) imagery CBM-I, (2) standard CBM-I (i.e., no instruction to use imagery), or (3) a neutral control condition. The participants will then practice their respective training at home for 7 days (60 scenarios/day). During this at-home training period, participants will track their worry three times per day. All the outcome measures will be reassessed at post-intervention, and 2-week follow-up. Worry will also be assessed at 1-week follow-up.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard cognitive bias modification (Experimental): Listen to descriptions of ambiguous scenarios that resolve positively
  Interventions: Behavioral: Standard cognitive bias modification
- Imagery enhanced cognitive bias modification (Experimental): Listen to descriptions of ambiguous scenarios that resolve positively while engaging in imagery
  Interventions: Behavioral: Imagery enhanced cognitive bias modification
- Neutral Control Condition (Placebo Comparator): Listen to descriptions of neutral scenarios
  Interventions: Behavioral: Neutral Control Condition

INTERVENTIONS:
Behavioral: Standard cognitive bias modification — Participants will be asked to repeatedly listen to descriptions of ambiguous scenarios that resolve positively and answer one question following each scenario that reinforces the positive interpretation; participants will listen to 60 scenarios/day for 7 days.
  Arms: Standard cognitive bias modification
Behavioral: Imagery enhanced cognitive bias modification — Participants will be asked to imagine themselves as though they are actively involved in the scenarios that they listen to. This condition will be required to answer two questions following each scenario; one that reinforces the positive interpretation and another that promotes engagement with imagery. Participants will listen to 60 scenarios/day for 7 days.
  Arms: Imagery enhanced cognitive bias modification
Behavioral: Neutral Control Condition — Participants will be asked to listen to descriptions of neutral (i.e., non-emotional) scenarios. This condition will also be required to answer one comprehension question following each scenario. Participants will listen to 60 scenarios/day for 7 days.
  Arms: Neutral Control Condition

SUMMARY:
People who experience high levels of worry often have mental habits that fuel their worry. One mental habit of interest to researchers is the tendency to assess situations and experiences in a very negative way even when it is possible the situation may turn out to be neutral or even positive. Cognitive bias modification of interpretations (CBM-I) is a training that is designed to target the tendency to catastrophize and jump to negative conclusions when faced with ambiguous information. CBM-I has been shown to improve this habit as well as anxiety and low mood. In this experiment, the investigators are looking to enhance CBM-I for pathological worry. Specifically, the investigators are testing the immediate and short-term effects of using imagery when completing CBM-I.

DETAILED DESCRIPTION:
In pathological worry, the tendency to assess situations and experiences in a very negative way even when it is possible the situation may turn out to be neutral or even positive is suggested to fuel worry. This type of "mental habit" can maintain worry and cause people a lot of distress. Cognitive bias modification of interpretations (CBM-I) involves repeatedly and actively listening to descriptions of ambiguous scenarios that resolve in a benign fashion. CBM-I has shown promise at reducing the tendency to make negative interpretations when presented with ambiguous information as well as improving worry and low mood. However, further research is needed to optimize the protocol for individuals who engage in pathological worry. One such way to improve the task is using imagery. In this proof-of-concept experiment, the investigators are looking at whether having participants use imagery while practicing CBM-I for one week leads to greater improvements in worry and worry-related processes compared to the standard protocol without imagery instructions and compared to a neutral control condition. This study will also investigate dosage effects of CBM-I training by investigating changes in worry over the intervention period using a daily diary assessment.

Potential participants will be asked to complete a telephone screen. Those who meet eligibility criteria will be invited to our laboratory at Ryerson University. After completing pre-intervention outcome measures, participants will be randomly assigned to one of three conditions: (1) a condition where people imagine themselves in scenarios they listen to; (2) a condition where people listen to the scenarios without instruction to use imagery; and (3) a condition in which people listen to passages of non-emotional situations. Participants will be asked to complete their respective training for 7 days (60 scenarios/day). There will be two follow-up visits; one after participants complete their training and another two weeks following completion of the training. All of the outcome measures will be assessed pre-intervention, post-intervention and at the 2-week follow-up. Past week worry will also be assessed at a 1-week follow-up via a link that will be emailed. During the 1-week intervention period participants will also track their worry 3 times per day via a link that will be emailed to them.

The present experiment will provide answers to important questions about the therapeutic potential of imagery enhanced CBM compared to standard CBM for pathological worry. Moreover, this study will shed light on dosing effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Score of 62 or higher on the Penn State Worry Questionnaire.
2. Endorsement of symptoms of Generalized Anxiety Disorder (e.g., excessive and uncontrollable worry) as per the DSM-5 description (American Psychiatric Association, 2013).

Exclusion Criteria:

1. Clinically significant suicidal ideation, intent, or plan
2. Past or current history of psychosis, bipolar disorder, or substance or alcohol use disorder over the past 12 months
3. Current psychological treatment or counseling unless this treatment is infrequent (once per month or less) or the participant has been receiving consistent weekly treatment for at least 12 weeks and still meets all other eligibility criteria
4. Psychotropic medication with a change in dose in the past 12 weeks. If they have recently discontinued a psychotropic medication, they will be included if it has been at least 1 month since discontinuation, or 3 months if they had been taking fluoxetine. Use of benzodiazepines in the past 12 weeks will also exclude participants.
5. Participants will be excluded if they report noncorrected hearing impairments as the training involves listening to audio recordings.
6. Participants will be excluded if they do not have daily access to a computer with internet as this is required to complete the at home training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported past-week worry as measured by the Penn State Worry Questionnaire-Past Week Version | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at 1-week and 2-week follow-ups.
  Self-report measure assessing the degree of excessive worry experienced over the past week. The measure contains 15 items and scores range from 0 to 90, with greater scores indicating a greater degree of worry.
Change in self-reported interpretation bias as measured by Ambiguous/ Unambiguous Situations Diary Extended | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at a 2-week follow-up.
  Self-report measure of interpretation bias that contains 55 vignettes describing a positive, negative, or ambiguous scenario. For each scenario, participants are instructed to rate their level of concern on a scale from 1 to 5, with higher scores indicating greater concern. Greater concern for ambiguous scenarios suggests greater interpretation bias.

SECONDARY OUTCOMES:
Self-reported depression, anxiety and stress as measured by the Depression, Anxiety and Stress Scale. | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at a 2-week follow-up.
  Self-report measure that assesses depression, anxiety and stress symptoms over the past week. The scale contains 21 items, divided into three subscales: 1) Depression, 2) Anxiety, and 3) Stress. Scores on the subscales range from 0 to 42, with higher scores indicating greater severity of depression, anxiety and stress.
Quality of problem solving as measured by the Means-Ends Problem-Solving task | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at a 2-week follow-up.
  Self-report measure of one's ability to conceptualize step-by-step strategies to solve two real-life problems. Problem solutions will be assessed for concreteness and effectiveness using a coding scheme.
Self-reported vividness, arousal, and likelihood of positive and negative prospective scenarios as measured by the Prospective Imagery Task | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at a 2-week follow-up.
  Self-report measure of the vividness and arousal associated with prospective positive and negative events, as well as the estimated likelihood that the prospective event might happen to them in the future. The scale contains 10 prospective positive events and 10 prospective negative events and ratings of vividness, arousal, and likelihood are made on a scale from 1 - 5, with higher scores indicating greater vividness, arousal, and likelihood.
Interpretation bias as measured by the Word-Sentence Association Paradigm | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at a 2-week follow-up.
  A computerized measure of interpretation bias. Participants are presented with an ambiguous sentence followed by a word that gives the sentence either a benign or threatening meaning. Participants are required to choose as quickly as possible whether the word is related to the ambiguous sentence (i.e., accept or reject). A greater tendency to 'accept' threatening interpretations and 'reject' benign interpretations would suggest a greater negative interpretation bias.
Self-reported negative thought intrusions as measured by the Breathing Focus Task | Administered on day 1 prior to completing the intervention (pre-intervention), following the intervention week (post-intervention), and at a 2-week follow-up.
  A behavioral measure of negative thought intrusions that involves a 5-minute breathing period, followed by a 5-minute period of instructed worry and then a second 5-minute breathing period. During the breathing periods, a tone sounds every 30 seconds and participants are instructed to report on whether they were focused on their breathing or if they had a thought intrusion. The thought intrusions are rated on their valence and the content of the intrusions is elaborated on further at the end of the task.
Daily Worry Questions | During the 7-day intervention period, all participants are asked to respond to questions about their worry three times per day (morning, afternoon, evening) using an online diary.
  A daily self-report measure of worry controllability, worry intensity, and distress associated with worry (all rated on a scale from 0 - 8) as well as time spent worrying (rated as a percentage).

OTHER OUTCOMES:
Self reported belief that the training will improve worry as measured by the Credibility Expectancy Check (CEQ) | Administered on day 1 prior to completing the intervention (pre-intervention) following the explanation of the intervention and the rationale.
  Self report measure assessing the extent to which the participant thinks and believes that the training will improve their worry. The measure has six questions in total; four questions are rated on a scale from 1 - 9 while the other two questions are rated on a scale from 0 - 100. Greater scores indicate greater expectations and perceptions of treatment credibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results of the study will be disseminated via conference presentations, journal publications, and through our lab website. Upon request, anonymized aggregate participant data may be made available to a publishing journal or individual research group. Individual research groups interested in accessing anonymized data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and CVs. Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal. No individual data will be shared.

REFERENCES:
- See also: Lab Website — https://psychlabs.ryerson.ca/caplab/